CLINICAL TRIAL: NCT00750932
Title: Study of the Biodistribution of PMN Serine Proteases in Sputum of Patients Affected by Cystic Fibrosis: Towards New Anti-inflammatory Therapies
Brief Title: Biodistribution of Neutrophile Proteases in the Sputum of Patients Affected by Cystic Fibrosis
Acronym: Pro-Muco
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: AOHP07-PD Pro-Muco; DGS2007-0295; N° ID RCB:2007-A00511-52; CPP: 2007-R17
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Sputum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- T: Control
- M: Minor with cystic fibrosis
- A: Adult with cystic fibrosis

SUMMARY:
The purpose of the proposed project is to characterize the neutrophile proteases which participate in the chronic inflammatory phenomenon associated with the cystic fibrosis and which are responsible for the degradation of the lung tissue.

The respiratory failure which results from it is one of main causes of the fatal evolution of this pathology but the anti-inflammatory therapies based on the use of antiproteases targeting specifically the soluble elastase did not end, until now, in the hoped results.

The identification of the other noxious targets is a crucial element to give new orientations to the anti-inflammatory strategies based on the administration of antiproteases which remain a promising way.

ELIGIBILITY:
Inclusion Criteria:

* Man /woman older than 18 years (for adult and group)
* Child aged 6 to 18 years (for child group)
* Suffering from cystic fibrosis in stable condition, ie not having presented thrust acute attack of the broncho-pulmonary or hospitalization for treatment of his illness during the previous 2 weeks

Exclusion Criteria:

* colonized by Burkholderia cepacia ou Stenotrophomonas maltophilia
* non smoker (control group)
* Without history or respiratory respiratory disease known (control group)
* Antibiotic treatment and / or anti-inflammatory drug (NSAID or corticosteroids) in the 2 weeks prior to the inclusion in the study (control group)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice DIOT, PHD, Principal Investigator — Tours Hospital
Locations (1):
- CHRU de Tours, Tours, France